CLINICAL TRIAL: NCT05551728
Title: Autism Caregiver Coaching in Africa
Acronym: ACACIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: University of Cape Town (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00111048
Record Dates: First submitted 2022-09-12; First posted 2022-09-23 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Autism or Autistic Traits
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Intervention Model Description: The study design will be an individually randomized group treatment RCT with a delayed treatment control group. 150 children, ages 18-72 months, with a DSM-5 diagnosis of autism spectrum disorder (ASD) and their caregivers will be recruited on a rolling basis, with arm allocation (coaching vs. delayed treatment control) conducted using a minimization approach with child sex balanced across groups. The intervention will be offered to the delayed treatment control group immediately after follow-up assessment (6-months after baseline). Offering the intervention to both groups is of ethical importance in an environment with few services and will enhance retention. Once control dyads have completed the intervention, the degree to which the trend in the control group is consistent with any treatment effect detected in the main trial comparison will be assessed. Note that a total of 320 participants will be enrolled in the study (150 caregiver-child dyads and 20 Aim 2 participants).
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, it is not possible to blind participants to the allocation received. Outcome assessors and statisticians will be blinded to participant group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): 12, 1-hour ESDM-informed caregiver coaching sessions, delivered by non-specialists. Intervention materials and approach have been adapted for the South African context.
  Interventions: Behavioral: ESDM-informed caregiver coaching
- Delayed intervention control group (No Intervention): Usual care.

INTERVENTIONS:
Behavioral: ESDM-informed caregiver coaching — The coaching intervention is informed by the Community-Early Start Denver Model (C-ESDM). The intervention has been adapted for the South African context. Training procedures have been adapted for delivery by non-specialist coaches. Twelve session-specific visuals with simple-text (for caregivers) and session scripts (for non-specialist coaches) have been developed. Over 12, 1-hour caregiver coaching sessions that are delivered by non-specialists, caregivers are coached in strategies to increase child attention to their social world, increase child communication, create and build joint activity routines, and understand and use the ABCs to support the development of new behaviors.
  Arms: Intervention group

SUMMARY:
Around the world there is a growing need to develop early intervention services in local communities that support a better quality of life for all autistic people. The South African study will test an approach where caregivers are coached by non-specialists in early intervention strategies. Caregivers can then use these strategies during everyday activities with their young autistic child.

DETAILED DESCRIPTION:
Globally there is a growing need to implement community-based services that support improvements in quality of life of autistic people. Early autism intervention is critical because it can significantly improve both child and family outcomes, but implementation gaps exist worldwide. These gaps are starkest in Africa, where by 2050, forty percent of the world's children will live. Given the lack of specialists in Africa, task shifting early autism intervention to non-specialists will be a key implementation strategy. Naturalistic Developmental Behavioral Interventions (NDBI), are a class of early autism intervention approaches, that can be effectively delivered by caregivers. Through a partnership between Duke University and the University of Cape Town, the team laid the groundwork for an innovative and scalable coaching intervention for young autistic children. A caregiver coaching NDBI was systematically adapted for the South African context in which coaching is effectively delivered by non-specialist Early Childhood Development practitioners employed by the Education Department. The proposed study will build on this foundational work by conducting a type 1 hybrid effectiveness implementation trial of the coaching intervention, delivered by non-specialists, within an existing system of care in South Africa. The goal is to implement a feasible, scalable early autism intervention model in Africa by conducting research with culturally and linguistically diverse participants in community-based settings, that is inclusive of diverse stakeholder perspectives and incorporates task-shifting. The proposed study will build on current relationships with families, practitioners, and policy makers by formalizing these relationships and including other key stakeholder groups such as South African autistic self-advocates through a community-academic partnership, a key bridging factor in the EPIS (Exploration, Preparation, Implementation, Sustainment) implementation framework. The proposed project has three main objectives. First, to evaluate the real-world effectiveness of non-specialist delivered NDBI caregiver coaching for improving patterns of caregiver-child interaction and child developmental outcomes, and assess the cost-effectiveness of this approach. Second, to identify implementation determinants to inform scale-up. Third, to expand African autism research capacity to enhance scalability. This project also offers a unique opportunity to study variability in autism-related behaviors and phenomenology. The study will therefore assess the degree to which response to intervention is moderated by caregiver and dimensional child characteristics. In addition, using an innovative digital assessment method, changes in dimensional quantitative measures of autism-related behaviors will be examined. Finally, cross-cultural differences in dimensional autism-related behaviors will be evaluated via comparison with existing quantitative phenotypic data gathered in U.S. studies. This study is timely and innovative and will inform scale-up of autism early intervention in Africa. Assessing the impact of a scalable intervention in an environment like South Africa which faces significant contextual challenges, increases the ecological validity and relevance of findings for many regions of the world that face with similar challenges.

ELIGIBILITY:
Inclusion Criteria:

* Child's age is 18-72 months
* Child meets DSM-5 criteria for autism spectrum disorder (ASD), informed by Autism Diagnostic Observation Schedule, Second Edition (ADOS-2)
* Child's caregiver speaks isiXhosa, isiZulu, Afrikaans, or English
* Child's race is African or Coloured (South African term for mixed race)
* Caregiver-child dyad live in recruitment area
* Caregiver is ≥18 years

Exclusion Criteria:

* Genetic disorder of known etiology (e.g., fragile X syndrome)
* Significant sensory or motor impairment that would preclude use of the play materials
* Major physical abnormalities that would interfere with participation in the intervention
* History of serious head injury and/or neurological disease
* Caregiver indicates they will be unable to attend assessments and 12 sessions

Ages: 18 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 320 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline VABS-3 Communication Domain Standard Score at 6 months | Baseline, 6 months
  The Vineland Adaptive Behavior Scales-3 (VABS-3) is a semi-structured, clinician-administered, caregiver interview that assesses the degree to which a child routinely performs specified adaptive behaviors compared to age-based norms, and yields standard scores for each subscale as well as an overall composite score. The measure examines domains of communication (receptive, expressive, and written language skills), socialization (play, interpersonal relationships, and coping skills),daily living skills (personal, domestic, and community living skills), and motor skills (gross and fine motor). Subscale score ranges from 20-140 where a higher score indicates greater frequency of target behavior.
Change from Baseline Griffiths III Language and Communication Developmental Quotient at 6 months | Baseline, 6 months
  The Griffiths Scales of Child Development, Third Edition (Griffiths III) is a comprehensive clinician-administered developmental measure designed for evaluation of children ranging in ages from birth to eight years. The Griffiths-III provides a profile of both strengths and weaknesses in child development across 5 domains: foundations of learning, language, and communication (expressive/receptive and social), eye and hand coordination (fine motor skills and visual perception), personal-social-emotional (emotional development and social interactions), and gross motor (postural control, balance, and body coordination). Developmental quotients (DQs) will be calculated by (Developmental Age/Chronological Age) *100, and range from 0-100 with higher scores indicating a higher degree of congruence between child developmental and chronological age.

SECONDARY OUTCOMES:
Change from Baseline JERI composite score at 4 months | Baseline, 4 months
  The Joint Engagement Rating Inventory (JERI) is a behavioral coding scheme designed to measure multiple aspects of caregiver-child interactions. The JERI includes 32 items rated on a 7-point Likert scale across four categories: 1) child engagement state items, 2) child activity items, 3) caregiver activity items, and 4) dyadic interaction items. For this study a JERI composite score will include the sum of 5 caregiver activity items including: scaffolding, following the child's interests, affect, language facilitation, and use of communicative temptations. Each caregiver activity item is rated on a 1-7 scale, with 1 indicating a low frequency and quality of the behavior and 7 indicating a high frequency and quality of the behavior.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cape Town, Cape Town, West Cape, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rieder AD, Viljoen M, Seris N, Shabalala N, Ndlovu M, Turner EL, Simmons R, de Vries PJ, Franz L. Improving access to early intervention for autism: findings from a proof-of-principle cascaded task-sharing naturalistic developmental behavioural intervention in South Africa. Child Adolesc Psychiatry Ment Health. 2023 May 20;17(1):64. doi: 10.1186/s13034-023-00611-0. PMID 37210513
- [Result] Franz L, Viljoen M, Askew S, Brown M, Dawson G, Di Martino JM, Sapiro G, Sebolai K, Seris N, Shabalala N, Stahmer A, Turner EL, de Vries PJ. Autism Caregiver Coaching in Africa (ACACIA): Protocol for a type 1-hybrid effectiveness-implementation trial. PLoS One. 2024 Jan 12;19(1):e0291883. doi: 10.1371/journal.pone.0291883. eCollection 2024. PMID 38215154
- [Result] Dawood Z, Sebolai K, Ndlovu M, Viljoen M, Seris N, Shabalala N, De Vries PJ, Franz L, Harty M. Detecting change in a caregiver-mediated autism intervention using the Joint Engagement Rating Inventory. S Afr J Commun Disord. 2025 Sep 26;72(1):e1-e11. doi: 10.4102/sajcd.v72i1.1102. PMID 41055175
- [Result] Viljoen M, Seris N, Shabalala N, Ndlovu M, de Vries PJ, Franz L. Adapting an early autism caregiver coaching intervention for telehealth delivery in low-resource settings: A South African study of the 'what' and the 'why'. Autism. 2025 May;29(5):1246-1262. doi: 10.1177/13623613241300774. Epub 2024 Dec 10. PMID 39655488